CLINICAL TRIAL: NCT00003165
Title: A Phase II Trial of PK1 in Women With Advanced Breast Cancer
Brief Title: Doxorubicin in Treating Women With Advanced Breast Cancer
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: University of Glasgow (Other)
Organization: National Cancer Institute (NCI) (NIH)
Purpose: Treatment
Other Study IDs: CDR0000065966; CRC-PHASE-II-PH2/038; EU-97028
Record Dates: First submitted 1999-11-01; First posted 2004-04-30 (Estimated); Last update posted 2013-12-19 (Estimated); Status verified 2010-04

CONDITIONS: Breast Cancer
Keywords: stage IV breast cancer; recurrent breast cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — doxorubicin-N-(2-hydroxypropyl)methacrylamide copolymer conjugate

INTERVENTIONS:
Drug: doxorubicin-HPMA conjugate

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die. Giving drugs in different forms may kill more tumor cells.

PURPOSE: Phase II trial to study the effectiveness of doxorubicin in treating women with advanced metastatic breast cancer.

DETAILED DESCRIPTION:
OBJECTIVES: I. Determine the antitumor activity of doxorubicin-HPMA conjugate (PK1) in women with advanced breast cancer.

OUTLINE: This is an open label, multicenter study. Patients receive doxorubicin-HPMA conjugate (PK1) by intravenous infusion once every 3 weeks. Patients may receive a total of 6 courses of treatment in the absence of toxicity and progressive disease.

PROJECTED ACCRUAL: 14-25 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS: Histologically or cytologically proven advanced metastatic carcinoma of the breast Bidimensionally measurable disease No brain or leptomeningeal disease

PATIENT CHARACTERISTICS: Age: Over 18 Performance status: WHO 0-2 Life expectancy: At least 3 months Hematopoietic: Hemoglobin at least 10 g/dL Neutrophil count at least 2,000/mm3 Platelet count at least 100,000/mm3 Hepatic: Bilirubin no greater than 11.7 mg/dL AST/ALT no greater than 2 times upper limit of normal (5 times upper limit of normal in presence of liver metastases) Renal: Creatinine no greater than 1.7 mg/dL Cardiovascular: No concurrent treatment for congestive cardiac failure Cardiac function within normal limits by MUGA or ECHO scan, if prior anthracycline therapy Other: Not pregnant or nursing Fertile patients must use effective contraception No concurrent nonmalignant systemic disease No active uncontrolled infection No prior history of malignant disease except: Squamous cell carcinoma of the skin Curatively treated carcinoma in situ of the cervix

PRIOR CONCURRENT THERAPY: Biologic therapy: No concurrent immunological therapy Chemotherapy: At least 1 prior chemotherapy regimen for advanced disease (including adjuvant therapy), but not more than 2 prior regimens At least 4 weeks since prior chemotherapy (6 weeks for nitrosourea or mitomycin) and recovered Cumulative dose of prior epirubicin no greater than 450 mg/m2 Cumulative dose of prior doxorubicin no greater than 240 mg/m2 No concurrent chemotherapy Endocrine therapy: No concurrent hormonal therapy Low dose steroid therapy allowed if dose established at least 4 weeks prior to study Radiotherapy: At least 4 weeks since prior radiotherapy and recovered Surgery: Not specified Other: No concurrent experimental therapy

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Estimated)
Dates: Start 1997-12

CONTACTS AND LOCATIONS:
Overall Officials: Chris Twelves, MD, BMedSci, FRCP, Study Chair — University of Glasgow
Locations (6):
- United Kingdom (6):
  - Cancer Research Campaign Clinical Trials Unit-Birmingham (CRCTU), Birmingham, England
  - Newcastle General Hospital, Newcastle upon Tyne, England
  - Weston Park Hospital, Sheffield, England
  - Aberdeen Royal Infirmary, Aberdeen, Scotland
  - Western General Hospital, Edinburgh, Scotland
  - Beatson Oncology Centre, Glasgow, Scotland